CLINICAL TRIAL: NCT03663608
Title: Wide Awake Local Anesthesia No Tourniquet
Acronym: WALANT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17-3065_WALANT
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Trigger Finger Disorder
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: WALANT Technique — pure local anaesthesia and without use of a tourniquet (WALANT Technique) for trigger finger release surger

SUMMARY:
The main objective is to assess patient's satisfaction regarding pure local anaesthesia and without use of a tourniquet (WALANT Technique) for trigger finger release surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age
* Isolated Trigger finger, diagnosis confirmed by sonography and with indication of surgical release
* Patients protected by health insurance
* Patients who have received proper information on the current research proctol, and did not refuse to enter the study

Exclusion Criteria:

* Hand vascular disorders ( History of finger replantation surgery, clinical signs of poor hand vascularization
* Hypersensitivy to Xylocain or Adrenalin or one of it's components
* Other surgical act planned to be performed during the same anaesthesia
* Pregnant or Breastfeeding women
* Patients of age and under the protection of a conservator, patients deprived of liberty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Isolated Trigger finger, diagnosis confirmed by sonography and indication of surgical release
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | one day after surgery
  Patient's agreement to use WALANT for possible surgeries to come and Patient's agreement to refer WALANT to his close relatives if they were to undergo surgery

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Privé de Plérin, Plérin
  - CHU de Rennes, Rennes